CLINICAL TRIAL: NCT01271218
Title: Effects of Glucosamine and Chondroitin Supplementation in Women With Knee Osteoarthritis Participating in an Exercise and Weight Loss Program: a Randomized Placebo Controlled Clinical Trial
Brief Title: Effects of Glucosamine and Chondroitin Supplementation in Women With Knee Osteoarthritis Participating in an Exercise and Weight Loss Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Baylor University (Other); Curves International (Industry)
Responsible Party: Richard B. Kreider, Department of Health & Kinesiology, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Curves-OA-06
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants ingested 2,200 mg/day of a placebo or active dietary supplement. Participants ingested three caplets in the morning and the remaining three caplets in the evening 30-minutes before a meal for 14-weeks. The supplements were prepared in caplet form and packaged in generic bottles for double blind administration. The placebo was a starch-based placebo matched for color, texture, and taste to the active supplement.
  Interventions: Other: Diet; Other: Exercise
- Active Supplement (Active Comparator): Participants were randomly assigned to ingest in a double-blind manner caplets containing a commercially available glucosamine/chondroitin (GC) dietary supplement (Curves Joint and Connective Support™, Curves International, Waco, TX) or a suitable placebo (P). The GC supplement provided a total of 1,500 mg/d of glucosamine, 1,200 mg/d of chondroitin sulfate, 120 mg/d of niacin, 120 mg/d of sodium, 45 mg/d of zinc, 900 mg/d MSM, 300 mg/d of boswellia serrata extract, 180 mg/d of white willow bark extract, and 15 mg/d of rutin powder. Participants ingested three caplets in the morning and the remaining three caplets in the evening 30-minutes before a meal for 14-weeks.
  Interventions: Other: Diet; Other: Exercise

INTERVENTIONS:
Other: Diet — Participants followed isoenergetic low fat diets with higher protein (HP) or higher carbohydrate (HC) macronutrient content. Participants consumed 1,200 kcals/d for 1-week (Phase I) and 1,600 kcals/d for 9-weeks (Phase II) during a 10-week weight loss period. Participants in the HC diet consumed a diet containing 55% carbohydrate, 15% protein, and 30% fat. Subjects in the HP group consumed a diet containing 7% carbohydrate, 63% protein, and 30% fat during Phase I of the diet and 15% carbohydrate, 55% protein, and 30% fat during Phase II of the diet. The final 4-weeks of the diet (Phase III) served as a weight maintenance period in which participants consumed 2,600 kcals•d-1 consisting of 55% carbohydrate, 15% protein, and 30% fat and were instructed to follow their respective Phase I diet (1,200 kcals/d) for 2-days only if they gained 1.35 kg (3 lbs).
  Other Names: Curves® weight loss program (Curves International, Waco, TX).
Other: Exercise — All subjects participated in a supervised exercise program three days per week for 14-weeks. Each circuit-style workout consisted of 14 exercises (e.g. elbow flexion/extension, knee flexion/extension, shoulder press/lat pull, hip abductor/adductor, chest press/seated row, horizontal leg press, squat, abdominal crunch/back extension, pec deck, oblique, shoulder shrug/dip, hip extension, side bends and stepping). Participants performed as many repetitions in a 30-s time period. In a continuous, interval fashion, participants performed floor-based callisthenic (e.g. running/skipping in place, arm circles, etc.) exercises on recovery pads for a 30-s time period after each resistance exercise in an effort to maintain a consistent exercise heart rate that corresponded to 60% to 80% of their maximum heart rate.
  Other Names: Curves exercise program.

SUMMARY:
Background: Exercise, weight loss, and dietary supplementation of glucosamine and chondroitin (GC) have been reported to improve functional capacity in individuals with knee osteoarthritis (OA). The purpose of this study was 1.) to determine whether women with knee OA who follow a higher protein diet observe more favorable changes in body composition and/or markers of health compared to those following a standard higher carbohydrate-based diet; and, 2.) to determine whether dietary supplementation of glucosamine and chondroitin during a weight loss and fitness program lessens symptoms of pain, improves functional capacity, and/or promotes greater health benefits in women with knee OA. It was hypothesized that both groups would experience beneficial changes in body mass, body composition, and markers of health. However, greater benefits would be observed in those following a higher protein diet while supplementing the diet with glucosamine and chondroitin.

DETAILED DESCRIPTION:
The study was conducted as a randomized, double-blind, placebo-controlled clinical trial in a university research setting. Participants with physician diagnosed OA participated in a 14-week fitness and weight loss program that consisted of moderately hypo-energetic higher protein or higher carbohydrate diets. Participants were also randomly assigned to ingest in a double-blind and randomized manner either a placebo or a commercially available dietary supplement containing glucosamine and chondroitin. Outcome measures were assessed at 0, 10, and 14 weeks of training, dieting, and supplementation.

ELIGIBILITY:
Inclusion Criteria:

- General entrance criteria included being a female with physician diagnosed OA between the ages of 18-70 years with a body mass index (BMI) > 27 kg/m2 and no recent participation in a diet or exercise program.

Exclusion Criteria:

- Subjects were not allowed to participate in this study if they: 1.) were pregnant, became pregnant, or had a desire for pregnancy; 2.) had any metabolic disorder including known electrolyte abnormalities, heart disease, arrhythmias, diabetes, thyroid disease, or hypogonadism; 3.) had a history of hypertension, hepatorenal, musculoskeletal, autoimmune, or neurological disease; were taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, or androgenic medications; 4.) had taken ergogenic levels of nutritional supplements that may affect muscle mass (e.g., creatine, HMB), anabolic/catabolic hormone levels (e.g., DHEA), or weight loss supplements (e.g., thermogenics) within three months prior to the start of the study; 5.) were ingesting any anti-inflammatory products two weeks before the start of the study or additional products during the study; 6.) reported any unusual adverse events associated with this study in which the supervising physician recommended removal from the study; 7.) had significant injury or surgery to the lower extremity or spine within the last six months; 8.) did not indicate a minimal amount of perceived pain and physical function limitation on inventories used in the study; 9.) had severe arthritis that required surgery and greatly limited functionality (inability to perform lunge); or, 10.) had arthritis that required the current use of physiotherapy modalities.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 14 weeks
  Perceptions of pain, knee flexibility, knee strength and endurance, upper body strength and endurance, peak aerobic capacity, and functional assessmentof balance using the sit to stand, step up and over, and forward lunge tests.

SECONDARY OUTCOMES:
Weight loss and body composition | 14 weeks
  All participants were tested for changes in energy intake; anthropometrics; body composition; and resting energy expenditure to assess magnitude of weight loss in response to a higher carbohydrate and higher protein diet.
Blood and Hormones | 14 Weeks
  General whole blood and serum clinical chemistries (cholesterol, triglycerides, glucose, blood urea nitrogen, creatinine, uric acid, muscle and liver enzymes) and hormones (C-Reactive Protein, IL-6, TNF-alpha, cortisol, insulin, homeostasis model of insulin sensitivity, and leptin).
Psychosocial | 14 Weeks
  SF-36 quality of life indices

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Exercise & Sport Nutrition Lab, College Station, Texas, United States

REFERENCES:
- [Derived] Magrans-Courtney T, Wilborn C, Rasmussen C, Ferreira M, Greenwood L, Campbell B, Kerksick CM, Nassar E, Li R, Iosia M, Cooke M, Dugan K, Willoughby D, Soliah L, Kreider RB. Effects of diet type and supplementation of glucosamine, chondroitin, and MSM on body composition, functional status, and markers of health in women with knee osteoarthritis initiating a resistance-based exercise and weight loss program. J Int Soc Sports Nutr. 2011 Jun 20;8(1):8. doi: 10.1186/1550-2783-8-8. PMID 21689421
- See also: Exercise & Sport Nutrition Lab — http://esnl.tamu.edu